CLINICAL TRIAL: NCT04989478
Title: Postprandial Metabolism in Healthy Young Subjects
Acronym: PoMet
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Bergen (Other)
Collaborators: Haukeland University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 236654
Record Dates: First submitted 2021-07-05; First posted 2021-08-04 (Actual); Last update posted 2022-01-06 (Actual); Status verified 2022-01

CONDITIONS: Postprandial Period; Biomarkers; Fasting
Keywords: Postprandial metabolism; Nutritional biomarker; Fasting
MeSH Terms: conditions — Fasting | interventions — Angptl4 protein, mouse

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Fasting — After the standardized breakfast meal, all participants will only consume water for 24 hours

SUMMARY:
This study aims to describe the dynamic changes in nutritional biomarkers in the blood during the postprandial period, i.e. the time period from the last meal and into the fasting state. In total 36 healthy, young men and women will be recruited in Bergen, Norway, and after receiving a standardized breakfast meal they will consume only water for the next 24 hours.

DETAILED DESCRIPTION:
Throughout the day, humans switch back and forth between the fed, postprandial (after a meal), and the postabsorptive (fasting) metabolic state. This is followed by a shift in fuel utilization from primarily using glucose to predominantly rely on β-oxidation of fatty acids. Consequently, circulating concentrations of biomarkers may fluctuate in response to this changing metabolic state. Much is known about the hormonal and metabolic effects of fasting, including lower insulin secretion, increased release of free fatty acids from adipose tissue, increased ketogenesis, glycogen breakdown, and activated gluconeogenesis. However, less is known about the effect on other biochemical markers in the postabsorptive period.

When evaluating nutritional biomarkers, both in clinical practice and in research, it is common practice to distinguish between fasting or non-fasting blood samples, based on time since the last meal. The extent to which different biomarkers are influenced by fasting status vary, and accordingly, several diagnostic cutoffs, e.g. plasma glucose for diabetes diagnosis, vary according to whether the sample was fasting or not. However, as the adaptation to fasting is a gradual process, it is expected that any changes in biomarker concentrations are also gradual. Further, as circulating metabolite concentrations are determined as a result of input (intestinal absorption and release from tissues), metabolism, and removal (utilization, storage, and excretion), we cannot reasonably assume that these changes are linear.

A few previous studies have aimed at describing the dynamics of fasting metabolism, demonstrating that the circulating metabolome changes during prolonged fasting in a dynamic manner. However, as data collection started after an overnight fast period, these studies do not provide data on the initial postprandial period and the adaptation to the fasting state. This study will extend the knowledge on the dynamics of human postprandial metabolism, by monitoring circulating concentrations of biomarkers during the 24 hours after a standardized breakfast meal. The investigators aim to capture the adaptation period from the fed to the fasting state and provide time-resolved data on a broad range of nutritional biomarkers.

Enrolled participants will attend the study center after an overnight fast, following a standardized evening meal consumed 12 hours before attendance. Anthropometric measurements (body weight, height, waist circumference, and body composition) will be taken in the fasting state, and a fasting blood sample will be drawn. After completing a standardized breakfast meal, the participants will remain at the study center for 12 hours, and blood will be frequently collected at specified time points. The participants will return to the study center the following morning for a final 24h fasting blood sample.

ELIGIBILITY:
Inclusion Criteria:

* Body Mass Index between 22-27 kg/m^2
* No significant weight change (>5%) during the last 3 months before the study visit
* Female participants should use one of the following oral contraceptives: Almina, Loette, Melleva, Microgynon, Mirabella, or Oralcon

Exclusion Criteria:

* Acute or chronic disease such as diabetes, thyroid diseases, cancer, cardiovascular disease, or inflammatory bowel disease, during the last 3 years
* Celiac disease or other food allergies interfering with the standardized breakfast meal
* Use of any prescription medications
* Smoking or regular use of other nicotine-containing products
* Pregnancy or breastfeeding the last 3 months

Ages: 20 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2021-08-16 (Actual); Primary Completion 2021-11-09 (Actual); Study Completion 2021-11-09 (Actual)

PRIMARY OUTCOMES:
Metabolomics profile in serum during 24 hour fasting | 24 hours
  Targeted metabolomics analyses of nutritional biomarkers related to B-vitamin status, one-carbon metabolism, and amino acids. All metabolite concentrations (Individual data + group geometric mean) will be presented for 14 prespecified timepoints after a standardized breakfast meal (15m, 30m, 45m, 60m, 90m, 2h, 3h, 4h, 6h. 8h, 10h, 12h, and 24h).

OTHER OUTCOMES:
Sex differences | 24 hours
  Comparison of metabolite concentrations between male and female subjects
Fasting vs nonfasting concentrations | 24 hours
  Comparison according to conventional cutoffs of fasting status (>6 and >8 hours)
12h fasting metabolomic profile after day vs night fast | 0 and 12 hours
  Compare 12h fasting concentrations after an overnight fast to 12h fasting concentrations after day fasting

CONTACTS AND LOCATIONS:
Locations (1):
- Research Unit for Health Surveys, University of Bergen, Bergen, Vestland, Norway

IPD SHARING:
Plan to Share IPD: Yes
Deidentified raw data will be deposited in a national research data repository (dataverse.no)
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: Immediately following publication. No end date.
Access Criteria: Anyone can access the data